CLINICAL TRIAL: NCT06602492
Title: Compensatory Behavior of E-cig Users in Response to Reduced Nicotine E-liquids
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rochester Institute of Technology (Other)
Responsible Party: Principal Investigator, Risa Robinson, Professor, Rochester Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21DA050852 (NIH)
Record Dates: First submitted 2024-09-15; First posted 2024-09-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy; Nicotine Addiction; Electronic Cigarette Use
Keywords: reduced nicotine eliquid; reduced exposure; cessation
MeSH Terms: conditions — Tobacco Use Disorder; Vaping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Switching Arm: High to Low Nicotine (Active Comparator): Baselined with a high nicotine eliquid and switched to a low nicotine eliquid.
  Interventions: Drug: Lower nicotine e-liquid
- Control Arm: High to High Nicotine (Placebo Comparator): Baselined with a high nicotine eliquid and continue with the same high nicotine eliquid.
  Interventions: Drug: Higher nicotine eliquid

INTERVENTIONS:
Drug: Lower nicotine e-liquid — A 3% nicotine concentration eliquid.
  Arms: Switching Arm: High to Low Nicotine
Drug: Higher nicotine eliquid — A 5% nicotine concentration eliquid.
  Arms: Control Arm: High to High Nicotine

SUMMARY:
The goal of this clinical trial is to learn if low nicotine eliquids work to reduce exposure to nicotine, in addicted ecig users, without increasing consumption of other harmful constituents.

The main questions it aims to answer are:

* Does switching to lower nicotine eliquids change the vaping behavior of addicted ecig users?
* Does switching to lower nicotine eliquids reduce the amount of nicotine consumed? Researchers will compare ecig users who switch from a higher to lower nicotine eliquid to a control group that does not switch.

Participants will:

* Complete history of tobacco use and nicotine addiction questionnaires
* Switch from higher to lower nicotine product or control for 15 days
* Complete daily questionnaires to report craving, mood and nicotine withdraw

For one full day under each nicotine condition, participants will:

* record puffing behavior using a topography monitor
* wear a sensorized shirt that measures the depth and duration of inhalation, and
* collect a saliva sample at the end of each day

DETAILED DESCRIPTION:
This project will investigate whether and how e-cig users compensate puff topography, lung inhalation, and cumulative consumption in response to reduced nicotine eliquid. The project is conducted in the natural environment to objectively measure if users adapt their behavior to maintain their desired level of nicotine.

The project employs a novel behavior-based exposure model that leverages the unique abilities of the investigative team to objectively capture real world behavior. The study employs a novel wPUM™ monitor to record puffing topography and a sensorized shirt to record respiratory parameters for every vaping session.

This study is conducted in the natural environment over 17 days. We will recruit N=80 current established adult ecig users, currently using eliquids with nicotine strengths greater than or equal to 5%, with no intention to quit e-cig use, and no use of combustible or other tobacco products. Participants will be randomized by age, gender, usual brand nicotine strength, and nicotine dependence score into a control arm (non-switching) and a test arm (switching). All participants will be baselined with 5% Juul ecigs and Juul pods containing Virginia Tobacco at 5% nicotine strength. The test arm will be switched to a 3% Juul pods containing Virginia Tobacco at 3% nicotine strength eliquid, while the control arm will continue to use 5% nicotine strength.

Participants will use the RIT wPUM monitor with a Juul ecig and a wearable sensorized garment to record their e-cigarette use topography and inhalation behavior ad-lib in their natural environment at the baseline and intervention conditions for one day each. Biosamples for nicotine exposure in saliva, NNAL in urine and CO will be collected, along with questionnaires to assess product use, compliance, and psychosocial outcomes such as craving, withdrawal and positive/negative emotional state.

Aim 1. Quantify changes in Total Particulate Matter (TPM) exposure among e-cig users adapting to low nicotine eliquids through compensatory changes in puffing, inhalation, and consumption behavior.

TPM exposure will be quantified in the natural environment by recording the topography (puff flow rate, duration, volume) of every puff taken along with respiratory behavior (inhalation/exhalation volume and time and breath hold). This novel outcome measure of exposure is used as a proxy to indicate the impact of behavior on increasing harm potential. We will test hypothesis (H1) that upon changing to a lower nicotine eliquid, users will adapt their behavior (i.e. increase breath hold, adjust puff flow rate, etc.), and in doing so will increase their TPM exposure.

Aim 2. Quantify changes in salivary among e-cig users adapting to low nicotine eliquids.

Salivary cotinine will be measured as a proxy to indicate efficacy of compensatory behavior. A Generalized Linear Mixed-Effects Model (GLME) analysis will be used to investigate how the ability of users to compensate for low nicotine e-liquids is affected by the presence of random effects including sex, age, nicotine dependence score, usual brand nicotine strength, and subjective effects including craving, withdrawal symptoms, and positive/negative emotional state. We will test the hypothesis (H2) that users are able to maintain desired nicotine levels while using a lower nicotine eliquid.

Relationship to Tobacco Regulation: Knowledge gained will support development of effective tobacco product regulations by informing three research questions of regulatory interest: (a) Will limiting the eliquid nicotine concentration reduce harm at the population level? (b) Is there evidence of compensatory behavior exhibited by e-cig users in response to reduced nicotine concentration, and (c) Can we conduct meaningful behavior-based e-cig use risk assessment at the individual level?

ELIGIBILITY:
Inclusion Criteria:

* 21 years or older
* Regular 30-day e-cig users

Exclusion Criteria:

* Intention to quit using e-cigs within the next 30 days
* Use of other tobacco products in addition to e-cigs on more than 9 of the previous 30 days
* History of acute or chronic asthma
* Previous diagnosis of cancer
* Other chronic medical conditions
* Use of chronic prescription medications
* Pneumonia in prior six weeks
* Upper respiratory tract infection or other febrile illness in previous 2 weeks
* Smokers on antioxidants, or anti-inflammatory therapy
* Pregnant women or women who intend to become pregnant or breast-feeding
* Had Covid-19 in the past 2 months or still feeling effects from a Covid-19 illness

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change in the Total Particular Mass (TPM) exposure when switching from the baseline to the intervention condition (high to low nicotine), based on the novel behavior-based yield model. | From enrollment to the end of 17 days.
  A behavior-based yield model, which combines product emissions with real-world user topography, is used to estimate the Change in Cumulative TPM exposure between low and high nicotine products.
  Total Particulate Mass (TPM) exposure of nicotine or other Harmful and Potentially Harmful Constituents (HPHCs) increases as a joint function of (1) the TPM delivered from the e-cig to the mouth, (2) the volume of diluting 'clean air' inhaled with the e-cig puff, and (3) the duration of time the emissions are in the lung.
  TPM exposure is proportional to the product of the TPM, which is the particulate mass contained in each puff delivered to the mouth (quantified by recording the volume of every puff and measuring the associated mass concentration in the emissions), v-inhale, which is the volume of air and entrained ecig aerosol inhaled into the lung with each puff (quantified with a senorized shirt), and t-cycle, which is the total time for the user to inhale each puff, hold their breath an

CONTACTS AND LOCATIONS:
Overall Officials: Risa J Robinson, PhD in Mechanical Engineering, Principal Investigator — Rochester Institute of Technology; Edward C Hensel, PhD in Mechanical Engineering, Study Director — Rochester Institute of Technology; Stephanie Godleski, PhD in Clinical Psychology, Study Director — Rochester Institute of Technology; Nathan Eddingsaas, PhD in Chemistry, Study Director — Rochester Institute of Technology
Locations (1):
- Rochester Institute of Technology, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No